CLINICAL TRIAL: NCT03470870
Title: Nomogram Control of Predictive Factors of Early Withdrawal After Gynecologic Oncology Surgery in the Enhanced Recovery After Surgery (ERAS) Protocol and Assessment of Practices
Acronym: NomogramGyneco
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: Nomogramme Gyneco-IPC 2017-034
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Gynecological Cancers
Keywords: Enhanced recovery after surgery; gynecologic oncology surgery; Nomogram control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients discharged before 2 days after surgery: patients discharged before 2 days of hospitalization following surgery
  Interventions: Other: Comparative analysis of the characteristics
- Patients discharged after 2 days after surgery: patients discharging after 2 days of hospitalization following surgery
  Interventions: Other: Comparative analysis of the characteristics

INTERVENTIONS:
Other: Comparative analysis of the characteristics — * Predictive nomogram of short-term hospitalization (less than two days after surgery)
  * Factors influencing the variations of average stay lenght
  * Morbidity of the ERAS program

SUMMARY:
Validation of a predictive nomogram of a short hospital stay (less than two days after surgery) on a prospective cohort of patients.

DETAILED DESCRIPTION:
* Validation of a predictive nomogram of short-term hospitalization (less than two days after surgery)
* Analysis of the factors influencing the variations of average length of stay
* Morbidity analysis of the ERAS program

ELIGIBILITY:
Inclusion Criteria:

* All patients who had surgery for gynecological cancer under the ERAS program.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had surgery for gynecological cancer under the RAAC program.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-01-08 (Estimated); Study Completion 2020-02-08 (Estimated)

PRIMARY OUTCOMES:
Validation of a predictive nomogram of a short hospital stay (less than two days after surgery) on a prospective cohort of patients. | 2 days
  Validation of a predictive nomogram of short-term hospitalization (less than two days after surgery)

SECONDARY OUTCOMES:
Descriptive analysis of the cohort. | 1 day
  Descriptive analysis of the cohort.
Analysis of the factors influencing the variations of average length of stay. | 1 day
  Analysis of the factors influencing the variations of the average duration of stay in time.
Analysis of the variation of the average duration of stay in time. | 1 day
  Analysis of the variation of the average duration of stay in time.
Morbidity analysis of the ERAS program. | 1 day
  Morbidity analysis of the ERAS program
Description of the implementation of the ERAS program on the entire cohort. | 1 day
  Description of the implementation of the ERAS program on the entire cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Eric LAMBAUDIE, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman JS, Roddy E, Ueda S, Brooks R, Chen LL, Chen LM. Enhanced Recovery Pathways for Improving Outcomes After Minimally Invasive Gynecologic Oncology Surgery. Obstet Gynecol. 2016 Jul;128(1):138-144. doi: 10.1097/AOG.0000000000001466. PMID 27275797
- [Background] Nicholson A, Lowe MC, Parker J, Lewis SR, Alderson P, Smith AF. Systematic review and meta-analysis of enhanced recovery programmes in surgical patients. Br J Surg. 2014 Feb;101(3):172-88. doi: 10.1002/bjs.9394. PMID 24469618
- [Background] Yoong W, Sivashanmugarajan V, Relph S, Bell A, Fajemirokun E, Davies T, Munro K, Chigwidden K, Evan F, Lodhi W; Enhanced Recovery After Surgery (ERAS) Team for Gynaecology and Anaesthesia. Can enhanced recovery pathways improve outcomes of vaginal hysterectomy? Cohort control study. J Minim Invasive Gynecol. 2014 Jan-Feb;21(1):83-9. doi: 10.1016/j.jmig.2013.06.007. Epub 2013 Jul 10. PMID 23850899
- [Background] Kroon UB, Radstrom M, Hjelthe C, Dahlin C, Kroon L. Fast-track hysterectomy: a randomised, controlled study. Eur J Obstet Gynecol Reprod Biol. 2010 Aug;151(2):203-7. doi: 10.1016/j.ejogrb.2010.04.001. Epub 2010 May 10. PMID 20452716
- [Background] Borendal Wodlin N, Nilsson L, Kjolhede P; GASPI study group. The impact of mode of anaesthesia on postoperative recovery from fast-track abdominal hysterectomy: a randomised clinical trial. BJOG. 2011 Feb;118(3):299-308. doi: 10.1111/j.1471-0528.2010.02697.x. Epub 2010 Sep 14. PMID 20840529
- [Background] Minig L, Chuang L, Patrono MG, Fernandez-Chereguini M, Cardenas-Rebollo JM, Biffi R. Clinical outcomes after fast-track care in women undergoing laparoscopic hysterectomy. Int J Gynaecol Obstet. 2015 Dec;131(3):301-4. doi: 10.1016/j.ijgo.2015.06.034. Epub 2015 Sep 8. PMID 26386495
- [Background] Bruneau L, Randet M, Evrard S, Damon A, Laurent FX. [Total laparoscopic hysterectomy and same-day discharge: Satisfaction evaluation and feasibility study]. J Gynecol Obstet Biol Reprod (Paris). 2015 Nov;44(9):870-6. doi: 10.1016/j.jgyn.2015.02.003. Epub 2015 Mar 13. French. PMID 25777619
- [Background] Chase DM, Lopez S, Nguyen C, Pugmire GA, Monk BJ. A clinical pathway for postoperative management and early patient discharge: does it work in gynecologic oncology? Am J Obstet Gynecol. 2008 Nov;199(5):541.e1-7. doi: 10.1016/j.ajog.2008.04.037. Epub 2008 Jun 2. PMID 18513685
- [Background] Wijk L, Franzen K, Ljungqvist O, Nilsson K. Enhanced Recovery after Surgery Protocol in Abdominal Hysterectomies for Malignant versus Benign Disease. Gynecol Obstet Invest. 2016;81(5):461-7. doi: 10.1159/000443396. Epub 2016 Jan 23. PMID 26799328
- [Background] Lindemann K, Kok PS, Stockler M, Jaaback K, Brand A. Enhanced Recovery After Surgery for Advanced Ovarian Cancer: A Systematic Review of Interventions Trialed. Int J Gynecol Cancer. 2017 Jul;27(6):1274-1282. doi: 10.1097/IGC.0000000000000981. PMID 28498237
- [Background] Vlug MS, Wind J, Hollmann MW, Ubbink DT, Cense HA, Engel AF, Gerhards MF, van Wagensveld BA, van der Zaag ES, van Geloven AA, Sprangers MA, Cuesta MA, Bemelman WA; LAFA study group. Laparoscopy in combination with fast track multimodal management is the best perioperative strategy in patients undergoing colonic surgery: a randomized clinical trial (LAFA-study). Ann Surg. 2011 Dec;254(6):868-75. doi: 10.1097/SLA.0b013e31821fd1ce. PMID 21597360
- [Background] Schlaerth AC, Abu-Rustum NR. Role of minimally invasive surgery in gynecologic cancers. Oncologist. 2006 Sep;11(8):895-901. doi: 10.1634/theoncologist.11-8-895. PMID 16951393
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Miralpeix E, Nick AM, Meyer LA, Cata J, Lasala J, Mena GE, Gottumukkala V, Iniesta-Donate M, Salvo G, Ramirez PT. A call for new standard of care in perioperative gynecologic oncology practice: Impact of enhanced recovery after surgery (ERAS) programs. Gynecol Oncol. 2016 May;141(2):371-378. doi: 10.1016/j.ygyno.2016.02.019. Epub 2016 Mar 9. PMID 26906066
- [Background] Kalogera E, Dowdy SC. Enhanced Recovery Pathway in Gynecologic Surgery: Improving Outcomes Through Evidence-Based Medicine. Obstet Gynecol Clin North Am. 2016 Sep;43(3):551-73. doi: 10.1016/j.ogc.2016.04.006. PMID 27521884
- [Background] Bauchat JR, Habib AS. Evidence-based anesthesia for major gynecologic surgery. Anesthesiol Clin. 2015 Mar;33(1):173-207. doi: 10.1016/j.anclin.2014.11.011. Epub 2014 Dec 31. PMID 25701935
- [Background] Touijer K, Scardino PT. Nomograms for staging, prognosis, and predicting treatment outcomes. Cancer. 2009 Jul 1;115(13 Suppl):3107-11. doi: 10.1002/cncr.24352. PMID 19544538
- [Background] Potters L, Roach M 3rd, Davis BJ, Stock RG, Ciezki JP, Zelefsky MJ, Stone NN, Fearn PA, Yu C, Shinohara K, Kattan MW. Postoperative nomogram predicting the 9-year probability of prostate cancer recurrence after permanent prostate brachytherapy using radiation dose as a prognostic variable. Int J Radiat Oncol Biol Phys. 2010 Mar 15;76(4):1061-5. doi: 10.1016/j.ijrobp.2009.03.031. Epub 2009 Jun 18. PMID 19540064
- [Background] Nixon IJ, Ganly I, Hann LE, Lin O, Yu C, Brandt S, Shah JP, Shaha A, Kattan MW, Patel SG. Nomogram for predicting malignancy in thyroid nodules using clinical, biochemical, ultrasonographic, and cytologic features. Surgery. 2010 Dec;148(6):1120-7; discussion 1127-8. doi: 10.1016/j.surg.2010.09.030. PMID 21134542
- [Background] Barsoum WK, Murray TG, Klika AK, Green K, Miniaci SL, Wells BJ, Kattan MW. Predicting patient discharge disposition after total joint arthroplasty in the United States. J Arthroplasty. 2010 Sep;25(6):885-92. doi: 10.1016/j.arth.2009.06.022. Epub 2009 Sep 2. PMID 19729270
- [Background] Kelly DM, Bennett R, Brown N, McCoy J, Boerner D, Yu C, Eghtesad B, Barsoum W, Fung JJ, Kattan MW. Predicting the discharge status after liver transplantation at a single center: a new approach for a new era. Liver Transpl. 2012 Jul;18(7):796-802. doi: 10.1002/lt.23434. PMID 22454258
- [Background] Wan KM, Carter J, Philp S. Predictors of early discharge after open gynecological surgery in the setting of an enhanced recovery after surgery protocol. J Obstet Gynaecol Res. 2016 Oct;42(10):1369-1374. doi: 10.1111/jog.13045. Epub 2016 Jun 29. PMID 27353883
- [Background] Schiavone MB, Herzog TJ, Ananth CV, Wilde ET, Lewin SN, Burke WM, Lu YS, Neugut AI, Hershman DL, Wright JD. Feasibility and economic impact of same-day discharge for women who undergo laparoscopic hysterectomy. Am J Obstet Gynecol. 2012 Nov;207(5):382.e1-9. doi: 10.1016/j.ajog.2012.09.014. Epub 2012 Sep 17. PMID 23107080